CLINICAL TRIAL: NCT06388499
Title: A Physiotherapy-led Disease-agnostic Telerehabilitation Programme for People With Chronic Health Conditions: a Mixed-methods Feasibility Trial
Brief Title: A Physiotherapy-led Disease-agnostic Telerehabilitation Programme for People With Chronic Health Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, RoisinCahalan, Associate Professor, University of Limerick
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIPG/2022/1854
Record Dates: First submitted 2024-04-19; First posted 2024-04-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Chronic Conditions, Multiple
Keywords: telerehabilitation; physiotherapy; feasibility; exercise; chronic conditions
MeSH Terms: conditions — Multiple Chronic Conditions; Motor Activity; Chronic Disease | interventions — Telerehabilitation; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TECC intervention group (Experimental): The intervention will comprise of a 6-week disease-agnostic exercise-based telerehabilitation programme for people with chronic health conditions delivered by a chartered physiotherapist. The intervention will consist of weekly synchronous exercise sessions and guided social component, and synchronous educational webinars to promote self-management of health and well-being. The intervention will be delivered remotely via telehealth. The intervention will include two exercise level groups (one seated class group conducting exercises in sitting, the other standing class conducting exercises in a range of standing/dynamic/functional positions). Allocation to the appropriate exercise level will be based on participants' baseline functional mobility level which will be assessed using the Activities-specific Balance Confidence (ABC) Scale.
  Interventions: Other: TECC (Telerehabilitation and Exercise for Chronic Conditions)

INTERVENTIONS:
Other: TECC (Telerehabilitation and Exercise for Chronic Conditions) — Exercise: Synchronous group exercise sessions will be delivered weekly via videoconferencing by a physiotherapist. Recordings of exercise sessions will be made available. Participants will be advised to perform additional exercise sessions at their own convenience to supplement the synchronous exercise sessions and facilitate adherence to physical activity guidelines.
  Education: A synchronous educational webinar will be delivered each week. These will be delivered by relevant healthcare professionals and explore various aspects of self-management of health and well-being. Recordings of the webinars will be made available to participants.
  Social component: At the end of each weekly synchronous group exercise session, participants will have the opportunity to engage in a 10-15-minute synchronous online social interaction with other participants in their exercise group via videoconferencing.

SUMMARY:
This protocol outlines a planned mixed methods feasibility trial which will be conducted to examine the feasibility and acceptability of a physiotherapy-led exercise-based telerehabilitation programme for groups of people with mixed chronic health conditions.

DETAILED DESCRIPTION:
Evidence supports the efficacy of exercise-based group rehabilitation programmes for people with chronic conditions. Telerehabilitation, referring to the remote delivery of rehabilitation using telecommunication technology, has the potential to increase service accessibility, uptake, and adherence to rehabilitation programmes. Telerehabilitation research has previously evaluated condition-specific programmes, such as cardiac telerehabilitation programmes delivered specifically to cardiac populations. However, recent evidence examining traditional in-person rehabilitation programmes points to the potential of rehabilitation programmes for mixed-condition patient groups as an efficient and pragmatic alternative approach to rehabilitation service delivery. The proposed study aims to examine the feasibility and acceptability of an exercise-based telerehabilitation programme delivered to groups of people with a mixture of different chronic conditions.

A mixed methods feasibility trial will be conducted to examine the feasibility of an exercise-based telerehabilitation programme for groups of people with mixed chronic health conditions. The 6-week intervention will involve exercise, educational, and social components. The intervention will include two different exercise group levels, one conducting a seat-based exercise class and the other a standing-based exercise class. Participants will take part in one synchronous group exercise session per week delivered via videoconferencing. This session will be followed by the opportunity to engage in a guided social discussion with peers via the videoconferencing platform. The social component of the intervention will be loosely structured and aims to provide a social dimension to the intervention, which has been previously identified by stakeholders as an important component of telerehabilitation programmes. The social discussion will be driven by patient preference and may refer to clinical issues such as supports or issues related to chronic conditions, or non-clinical issues related to current news/events. Participants will be provided access to a synchronous online self-management educational webinar each week also delivered via videoconferencing. Access to recordings of the exercise classes and educational webinars will also be provided to allow participants to engage with the sessions at their convenience during the intervention period. Data will be collected and analysed to address outcomes of feasibility and acceptability including recruitment, retention, intervention adherence including adherence with synchronous exercise and education sessions and with recorded exercise and education content, participant satisfaction, safety, participant experiences and clinical effectiveness of the intervention.

The proposed feasibility trial will guide new iterations and evaluation and potentially a future definitive randomised control trial evaluating the use of exercise-based telerehabilitation interventions for groups of people with mixed chronic health conditions. The proposed intervention has been designed with the aim of developing a sustainable, cost-effective, and efficacious healthcare delivery method to tackle the increasing demand for rehabilitation programmes for people with chronic health conditions.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults (aged ≥18 years old) with a confirmed diagnosis of any chronic cardiorespiratory, neurological, or musculoskeletal condition. We will use the ICD-10-CM definition of a chronic condition being one lasting greater than 12 months and resulting in the need for ongoing medical intervention and limiting self-care, independent living, and social interaction.
* Person is medically stable and appropriate to participate in the exercise-based intervention independently and safely as deemed by self-declaration. Participants who fulfil the criteria will undergo screening by the research team to gather relevant medical history and will be required complete the Physical Activity Readiness Questionnaire (PAR-Q) form. If any concerns arise from the PAR-Q form, participants will be advised to discuss their suitability for participation in the intervention with their GP in advance of signing the disclaimer prior to participation. Participants will be required to sign a disclaimer to agree voluntary participation in the exercise intervention at their own risk prior to participating.
* Access to an appropriate technological device with an internet connection and email address to facilitate participation in the telerehabilitation intervention.
* Willing to provide informed consent to participate in the study.
* Good level of spoken and written English.

Exclusion Criteria:

* Adults who are medically unstable as deemed by referring physiotherapist or who have uncontrolled medical conditions limiting participation in exercise interventions including uncontrolled hypertension or recent acute cardiovascular events, uncontrolled atrial fibrillation, etc.
* Significant orthopaedic, psychological, neurological, or cognitive conditions or mobility difficulties that prevents participation in seated or standing exercise interventions as deemed by referring physiotherapist.
* Suspected underlying malignancy as deemed by referring physiotherapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Recruitment rate assessed by number of participants recruited during recruitment period. | 4 weeks
  The number of participants recruited over a 4-week recruitment period
Retention rate assessed by the proportion of enrolled participants who complete post-intervention assessments. | 8 weeks
  The percentage of enrolled participants who complete the post-intervention assessments and focus groups
Adherence rate assessed by the attendance at synchronous group exercise sessions | 6 weeks
  Adherence with the overall intervention will be recorded by the attendance of participants at the synchronous group exercise sessions throughout the 6-week intervention period which will be recorded by the researchers.
Satisfaction with the intervention as assessed by the Client-Satisfaction Questionnaire 8 (CSQ-8) | 6 weeks
  Satisfaction with the overall intervention will be examined using the Client-Satisfaction Questionnaire 8 (CSQ-8). The CSQ-8 scale is an 8-item scale which rates satisfaction on a 4-point Likert scale. An overall score is calculated by summing the respondent's rating score for each scale item with totals ranging from 8 to 32, with higher values indicating higher satisfaction
Satisfaction with individual intervention components assessed by Numerical Rating Scales (NRS) | 6 weeks
  Participant satisfaction with individual components of the intervention (including the orientation session, exercise sessions, educational webinars, and social components) will be assessed using Numerical Rating Scales (NRS).
Adverse events assessed via self-report questionnaire | 6 weeks
  Participants will be asked during the post-intervention assessment to report the occurrence of any adverse events during the intervention period via a custom questionnaire. Adverse events will be defined as any problems or injuries experienced during the study that is deemed by the participant to be more likely resulting from participation in the intervention, rather than resulting from disease progression. Serious adverse events will be defined as any medical occurrence resulting in death, threat to life, hospital admission or significant disability.
Intervention acceptability as assessed by qualitative feedback from participants via focus groups | 6 weeks
  Qualitative semi-structured focus groups will be carried out to collect data regarding patient experiences and acceptability of the intervention.

SECONDARY OUTCOMES:
Physical function assessed by the 30-second chair stand test (30CST). | 6 weeks
  The 30-second chair stand test (30CST) will be administered both pre-intervention and post-intervention to assess the effect of the intervention on objective physical function.
Quality of life assessed by the Euro-QoL 5 Dimension 5 Level (Euro-QoL-5D-5L). | 6 weeks
  The Euro-QoL 5 Dimension 5 Level (Euro-QoL-5D-5L) will be administered in pre-intervention and post-intervention assessments to assess the effect of the intervention on quality of life. The Euro-QoL-5D-5L is a patient-reported outcome measure which assesses health-related quality of life across five dimensions of health using a 5-point rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Roisin Cahalan, PhD, Principal Investigator — University of Limerick, Ireland
Locations (1):
- South Tipperary Chronic Disease Management Hub, St. Brigid's Hospital, Carrick-on-Suir, Tipperary, Ireland